CLINICAL TRIAL: NCT02262988
Title: Thigh Pain After Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondren Orthopedic Group L.L.P. (Other)
Collaborators: InGeneron, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOG-TOH175
Record Dates: First submitted 2014-09-30; First posted 2014-10-13 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
Keywords: knee; joint replacement; total knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tourniquet used with intramedullary rod (Experimental): Patients will undergo a total knee replacement with a tourniquet and intramedullary rod.
  Interventions: Procedure: Total knee replacement
- No tourniquet with intramedullary rod (Experimental): Patients will undergo a total knee replacement without a tourniquet and with an intramedullary rod.
  Interventions: Procedure: Total knee replacement
- Tourniquet without intramedullary rod (Experimental): Patients will undergo a total knee replacement with a tourniquet and without an intramedullary rod.
  Interventions: Procedure: Total knee replacement
- No tourniquet without intramedullary rod (Experimental): Patients will undergo a total knee replacement without a tourniquet nor an intramedullary rod.
  Interventions: Procedure: Total knee replacement

INTERVENTIONS:
Procedure: Total knee replacement — Total knee replacement (TKA)

SUMMARY:
The purpose of this research study is to evaluate the cause of thigh pain after knee replacement. Different surgical techniques will be used to help determine the cause of thigh pain, and all surgical techniques are accepted and produce good clinical results.

DETAILED DESCRIPTION:
This research study will be a randomized study in which patients volunteer participate. "Randomized" means the patients who received the new treatment are chosen at random, similar to flipping a coin. Several factors have been identified as possible sources of thigh pain after surgery: use of a tourniquet around the thigh to control bleeding during surgery; use of an intramedullary rod during surgery or quadriceps muscle strain. Participants will be randomized into surgical groups that use/do not use a tourniquet and use/do not use intramedullary rod during surgery. A subset of participants in all surgical groups will have a MRI to look for quadriceps muscle strain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing total knee arthroplasty for osteoarthritis
* Adult patients (age 18 years or older)
* Written informed consent
* Ability to speak, read and write English or Spanish

Exclusion Criteria:

* Inability to speak, read and write English or Spanish
* Evidence of malignant disorder/neoplasm in past 60 months
* Contraindication for removal of infrapatellar fat pad
* History of smoking and not committed to give up
* Chronic skin conditions
* Connective, metabolic or skin disease
* Evidence of active infection
* Pregnancy or lactating for female subjects
* Current corticosteroid use
* Immunosuppressive medication
* Renal failure (creatine > 1.8 mg/dL)
* Hepatic failure (AST, ALT > 2x normal values; bilirubin > 2 mg/dL)
* Inflammatory joint diseases of the knee that indicate additional, conflating therapies
* Joint infection within the past 6 months
* No prisoners or mentally disabled persons
* No Workers' Compensation cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Survey (KOOS) | up to 3 months
  Survey

SECONDARY OUTCOMES:
Pain Scores on Numerical Rating Scale | up to 3 months
  Pain scale from 0-10 with 0 representing no pain and 10 representing maximum pain.
Knee swelling | up to 3 months
  Physician evaluation
Knee Range of Motion | up to 3 months
  Goniometer measurement
Number of Patients with Adverse Events as a Measure of Safety | up to 3 months
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gregory W Stocks, MD, Principal Investigator — Fondren Orthopedic Group L.L.P.
Locations (1):
- Fondren Orthopedic Group, L.L.P., Houston, Texas, United States